CLINICAL TRIAL: NCT07166627
Title: Surgical Excision Versus Ultrasound Guided Evacuation of Cesarean Section Scar Ectopic Pregnancy Type II: A Comparative Study
Brief Title: Comparison Between Surgical Excision and Ultrasound Guided Evacuation in Management of Cesarean Section Scar Pregnancy.
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Fahmy, specialist of OB/GYN, Sohag University
Other Study IDs: Soh-Med-25-8-6MD
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Scar Pregnancy
Keywords: cesarean scar pregnancy; evacuation of CSP; surgical excision of CSP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ultrasound guided evacuation
  Interventions: Procedure: ultrasound guided evacuation of cesarean section scar ectopic pregnancy
- surgical excision
  Interventions: Procedure: surgical excision of cesarean section scar ectopic pregnancy

INTERVENTIONS:
Procedure: surgical excision of cesarean section scar ectopic pregnancy — surgical excision by laparotomy.
  Groups: surgical excision
Procedure: ultrasound guided evacuation of cesarean section scar ectopic pregnancy — ultrasound guided evacuation of cesarean section scar ectopic pregnancy trans-cervically.
  Groups: ultrasound guided evacuation

SUMMARY:
patients diagnosed with cesarean section scar ectopic pregnancy type II will be divided into two groups, one will undergo surgical excision and the other one will undergo ultrasound-guided evacuation in order to compare safety and efficacy of both techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with cesarean scar ectopic pregnancy Type II in the 1st trimester.

Exclusion Criteria:

* patients with cesarean scar pregnancy type 2 above 14 weeks.
* Type I and type III cesarean section scar pregnancy.
* patients presented with massive bleeding or shock.
* Heterotopic pregnancy.
* Simultaneous Hysterectomy or Sterilization.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: patients diagnosed with cesarean section scar ectopic pregnancy type II and undergoing treatment in sohag university hospital.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of surgical excision versus ultrasound guided evacuation of cesarean section scar ectopic pregnancy. | 1 year

SECONDARY OUTCOMES:
hematoma formation | 1 year
bleeding above 1 liter | 1 year
recurrence of cesarean section scar ectopic | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hazem M Mohamed, MD, Study Chair — Sohag University; Mohamed N Salem, MD, Study Director — Sohag University; Mohammed S Ismail, MD, Study Director — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No